CLINICAL TRIAL: NCT07330323
Title: Development and Evaluation of a Personalized Discharge Letter for Low-risk Skin Cancer Patients After Dermatological Screening.
Brief Title: CARES : Customized Aftercare Report for Evaluated Skin Cancer Patients
Acronym: CARES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S70829
Record Dates: First submitted 2025-12-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Management; Low Risk; Skin Cancer
Keywords: Skin cancer risk and management; personalized discharge letter; low-risk skin cancer patients
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Standard of Care (Active Comparator): Verbal information only.
  Interventions: Behavioral: Verbal information only
- Group B: Personalized Discharge Letter (Experimental): Tailored written information based on individual risk profile, skin type and consultation findings.
  Interventions: Behavioral: Personalized Discharge Letter
- Group C: Personalized Discharge Letter + Digital Visual Support (IntelliStudio) (Experimental): Tailored written information plus digital visual support (e.g. annotated images, visual summaries).
  Interventions: Behavioral: Personalized Discharge Letter + IntelliStudio

INTERVENTIONS:
Behavioral: Verbal information only — Verbal information only
  Arms: Group A: Standard of Care
Behavioral: Personalized Discharge Letter — Personalized Discharge Letter: Tailored written information based on individual risk profile, skin type and consultation findings.
  Arms: Group B: Personalized Discharge Letter
Behavioral: Personalized Discharge Letter + IntelliStudio — Personalized Discharge Letter + IntelliStudio: Tailored written information plus digital visual support (e.g. annotated images, visual summaries).
  Arms: Group C: Personalized Discharge Letter + Digital Visual Support (IntelliStudio)

SUMMARY:
Current clinical practices often provide general verbal advice to low-risk patients, which may not sufficiently address individual concerns or offer actionable steps. Generic information on the internet can be overwhelming or unreliable, leading to confusion and unnecessary follow-up visits.

This project introduces a tailored approach by combining evidence-based guidelines with personalized details about the patient's risk profile. The discharge letter bridges the gap between clinical expertise and patient understanding, offering clear, specific, and actionable advice that has been shown to improve health behaviors and outcomes in other contexts .

The personalized discharge letters are generated using an AI agent trained on validated letters from the hospital's electronic health record system (KWS). Each letter is reviewed and approved by a physician before being provided to the patient, ensuring both accuracy and clinical relevance.

DETAILED DESCRIPTION:
This study is a prospective, parallel-group, open-label, randomized controlled trial designed to evaluate the impact of a personalized discharge letter-with or without digital visual support -on reassurance, knowledge, and self-management in low-risk skin cancer patients following dermatological screening.

Study Arms: Participants will be randomly assigned to one of three groups:

* Group A - Standard of Care: Verbal information only.
* Group B - Personalized Discharge Letter: Tailored written information based on individual risk profile, skin type and consultation findings.
* Group C - Personalized Discharge Letter + digital visual support: Tailored written information plus digital visual support (e.g. annotated images, visual summaries).

Scientific Rationale Current discharge practices for low-risk skin cancer patients often rely on general verbal advice, which may not sufficiently address individual concerns or promote long-term self-care. Evidence from other medical domains suggests that personalized communication improves patient understanding, satisfaction, and adherence to follow-up recommendations.

This study introduces an AI agent trained on validated discharge letters from the hospital's electronic health record system (KWS). The AI helpt collect information from the electronic health record that is relevant for creating personalized letters that are reviewed by a physician before being provided to the patient. These letters aim to improve understanding of personal skin cancer risk, sun protection, and self-monitoring practices.

The addition of visual digital support (IntelliStudio) is hypothesized to further enhance patient engagement and confidence by providing clear, visual explanations of findings and next steps. This design allows for a direct comparison of standard care versus increasingly personalized interventions, enabling the evaluation of both individual and combined effects.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Low-risk skin cancer patients:

  1. Negative personal history for melanoma
  2. Less than 100 naevi
  3. Less than 5 clinically atypical naevi
  4. Maximum 1 BCC in history
  5. Maximum 1 SCC, and at least 5 years ago
  6. AK: treated and controlled with clinical response
  7. M Bowen: treated and controlled with clinical response
* Adult subjects (between 18 years of age and 80 years) at time of enrolment

Exclusion Criteria:

* Presence of dermatological lesions requiring immediate treatment at the time of consultation.
* History of solid organ transplantation (Organ Transplant Recipient, OTR).
* Known carriers or suspected carriers (based on family history) of germline mutations associated with increased skin cancer risk (e.g. CDKN2A, PTCH1, XP genes).
* Failure to meet one or more of the inclusion criteria.
* Any condition or comorbidity that, in the opinion of the investigator, may interfere with study participation or data interpretation (e.g. severe cognitive impairment, language barrier).
* Participation in another interventional clinical trial that may interfere with the outcomes of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Level of Reassurance Immediately Post-Consultation | Through study completion, an average of 1 year
  Measured via a questionnaire.
  Hypothesis: Patients in the IntelliStudio group will report the highest levels of reassurance.
Knowledge of Personal Skin Cancer Risk | Through study completion, an average of 1 year
  Assessed through a pre- and post-intervention knowledge questionnaire.
  Hypothesis: Personalized information (Groups B and C) improves risk awareness compared to standard care.
Confidence in Performing Self-Skin Checks | Through study completion, an average of 1 year
  Measured via self-reported confidence and frequency of self-checks.
  Hypothesis: Groups B and C will report higher confidence than Group A.

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Department of Dermatology, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No